CLINICAL TRIAL: NCT00439296
Title: A Phase I/II Trial of ABT-751 Combined With Dexamethasone, PEG-asparaginase, and Doxorubicin in Relapsed Acute Lymphoblastic Leukemia (ALL)
Brief Title: ABT-751 With Chemotherapy for Relapsed Pediatric ALL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to poor accrual and lack of funding.
Sponsor: Therapeutic Advances in Childhood Leukemia Consortium (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: T2005-001
Record Dates: First submitted 2007-02-21; First posted 2007-02-23 (Estimated); Results first posted 2020-09-09 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-02

CONDITIONS: Recurrent Pediatric ALL; Relapsed Pediatric ALL; Acute Lymphoblastic Leukemia; Refractory Pediatric ALL
Keywords: Acute Lymphoblastic Leukemia; Pediatrics; Relapsed; Recurrence; ABT-751; Therapeutic Advances in Childhood Leukemia; Investigational; Childhood; ALL; Relapsed ALL; Refractory ALL; Relapsed pediatric ALL; Refractory pediatric ALL; TACL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence | interventions — ABT751; Antineoplastic Agents; Dexamethasone; Calcium Dobesilate; pegaspargase; Asparaginase; asparaginase erwinia chrysanthemi recombinant; Doxorubicin; Cytarabine; Methotrexate; Cyclophosphamide; Thioguanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Dose Level 1 (Experimental): Treatment Dose of ABT-751 is 80 mg/m2/day
  Tx Course 1:
  • ABT-751, Dexamethasone, PEG-asparaginase, Doxorubicin, Cytarabine, IT Methotrexate
  Tx Course 2:
  • Cyclophosphamide, 6-Thioguanine, IT Methotrexate, Cytarabine, PEG-asparaginase, ABT-751
  Tx Courses 3-12 (maintenance courses):
  • ABT-751, IT Methotrexate
  Interventions: Drug: ABT-751; Drug: Dexamethasone; Drug: PEG-asparaginase; Drug: Doxorubicin; Drug: Cytarabine; Drug: Methotrexate; Drug: Cyclophosphamide; Drug: 6-thioguanine
- Dose Level 2 (Experimental): Treatment Dose of ABT-751 is 100 mg/m2/day
  Tx Course 1:
  • ABT-751, Dexamethasone, PEG-asparaginase, Doxorubicin, Cytarabine, IT Methotrexate
  Tx Course 2:
  • Cyclophosphamide, 6-Thioguanine, IT Methotrexate, Cytarabine, PEG-asparaginase, ABT-751
  Tx Courses 3-12 (maintenance courses):
  • ABT-751, IT Methotrexate
  Interventions: Drug: ABT-751; Drug: Dexamethasone; Drug: PEG-asparaginase; Drug: Doxorubicin; Drug: Cytarabine; Drug: Methotrexate; Drug: Cyclophosphamide; Drug: 6-thioguanine
- Dose Level 3 (Experimental): Treatment Dose of ABT-751 is 125 mg/m2/day
  Tx Course 1:
  • ABT-751, Dexamethasone, PEG-asparaginase, Doxorubicin, Cytarabine, IT Methotrexate
  Tx Course 2:
  • Cyclophosphamide, 6-Thioguanine, IT Methotrexate, Cytarabine, PEG-asparaginase, ABT-751
  Tx Courses 3-12 (maintenance courses):
  • ABT-751, IT Methotrexate
  Interventions: Drug: ABT-751; Drug: Dexamethasone; Drug: PEG-asparaginase; Drug: Doxorubicin; Drug: Cytarabine; Drug: Methotrexate; Drug: Cyclophosphamide; Drug: 6-thioguanine
- Dose Level 4 (Experimental): Treatment Dose of ABT-751 is 150 mg/m2/day
  Tx Course 1:
  • ABT-751, Dexamethasone, PEG-asparaginase, Doxorubicin, Cytarabine, IT Methotrexate
  Tx Course 2:
  • Cyclophosphamide, 6-Thioguanine, IT Methotrexate, Cytarabine, PEG-asparaginase, ABT-751
  Tx Courses 3-12 (maintenance courses):
  • ABT-751, IT Methotrexate
  Interventions: Drug: ABT-751; Drug: Dexamethasone; Drug: PEG-asparaginase; Drug: Doxorubicin; Drug: Cytarabine; Drug: Methotrexate; Drug: Cyclophosphamide; Drug: 6-thioguanine
- Dose Level 5 (Experimental): Treatment Dose of ABT-751 is 175 mg/m2/day
  Tx Course 1:
  • ABT-751, Dexamethasone, PEG-asparaginase, Doxorubicin, Cytarabine, IT Methotrexate
  Tx Course 2:
  • Cyclophosphamide, 6-Thioguanine, IT Methotrexate, Cytarabine, PEG-asparaginase, ABT-751
  Tx Courses 3-12 (maintenance courses):
  • ABT-751, IT Methotrexate
  Interventions: Drug: ABT-751; Drug: Dexamethasone; Drug: PEG-asparaginase; Drug: Doxorubicin; Drug: Cytarabine; Drug: Methotrexate; Drug: Cyclophosphamide; Drug: 6-thioguanine
- Dose Level 0 (Experimental): Treatment Dose of ABT-751 is 65 mg/m2/day
  Tx Course 1:
  • ABT-751, Dexamethasone, PEG-asparaginase, Doxorubicin, Cytarabine, IT Methotrexate
  Tx Course 2:
  • Cyclophosphamide, 6-Thioguanine, IT Methotrexate, Cytarabine, PEG-asparaginase, ABT-751
  Tx Courses 3-12 (maintenance courses):
  • ABT-751, IT Methotrexate
  Interventions: Drug: ABT-751; Drug: Dexamethasone; Drug: PEG-asparaginase; Drug: Doxorubicin; Drug: Cytarabine; Drug: Methotrexate; Drug: Cyclophosphamide; Drug: 6-thioguanine
- Dose Level -1 (Experimental): Treatment Dose of ABT-751 is 50 mg/m2/day
  Tx Course 1:
  • ABT-751, Dexamethasone, PEG-asparaginase, Doxorubicin, Cytarabine, IT Methotrexate
  Tx Course 2:
  • Cyclophosphamide, 6-Thioguanine, IT Methotrexate, Cytarabine, PEG-asparaginase, ABT-751
  Tx Courses 3-12 (maintenance courses):
  • ABT-751, IT Methotrexate
  Interventions: Drug: ABT-751; Drug: Dexamethasone; Drug: PEG-asparaginase; Drug: Doxorubicin; Drug: Cytarabine; Drug: Methotrexate; Drug: Cyclophosphamide; Drug: 6-thioguanine

INTERVENTIONS:
Drug: ABT-751 — Treatment Course 1:
  Oral capsule to be given daily for 21 days at assigned dose.
  Treatment Course 2:
  ABT-751 will be taken once daily, by mouth, at the assigned dose on days 15-35.
  Treatment Course 3:
  ABT-751 will be taken once daily, by mouth, at the assigned dose on days 1-21 followed by 1 week of rest.
  Other Names: Antineoplastics
Drug: Dexamethasone — In Treatment Course 1 only:
  * 10 mg/m2/day divided BID.
  * Take dexamethasone by mouth days 1-14.
  Other Names: Decadron; Dexasone; Diodex; Hexadrol; Maxidex
Drug: PEG-asparaginase — In Treatment Course 1:
  * 2500 IU's/m2/day.
  * Intramuscular injection (IM) on days 4, 11 and 18.
  In Treatment Course 2:
  * 2500 IU's/m2/day.
  * Intramuscular injection (IM) on day 15.
  Other Names: Elspar; Kidrolase; L-asparaginase; Erwinia L-asparaginase
Drug: Doxorubicin — In Treatment Course 1 only:
  • 60 mg/m2/day IV over 15 minutes on day 1.
  Other Names: Adriamycin; Rubex
Drug: Cytarabine — * Given Intrathecally on day 1 of course 1 at the dose defined by age below.
    * 30 mg for patients age 1-1.99
    * 50 mg for patients age 2-2.99
    * 70 mg for patients >3 years of age
  * Omit IT Ara-C on Day 1 if patient received IT therapy prior to study enrollment as part of diagnostic lumbar puncture procedure.
  In Treatment Course 2: • 75 mg/m2/day IV on days 2 through 5 and days 9 through 12.
  Other Names: Cytosar-U; Ara-C; Arabinosylcytosine
Drug: Methotrexate — In Treatment Course 1:
  • Given Intrathecally on day 15 at the dose defined by age below.
  * 8 mg for patients age 1-1.99
  * 10 mg for patients age 2-2.99
  * 12 mg for patients 3-8.99 years of age
  * 15 mg for patients >9 years of age
  In Treatment Course 2:
  • Given Intrathecally on day 1, 8, 15 and 22 at the dose defined by age below.
  * 8 mg for patients age 1-1.99
  * 10 mg for patients age 2-2.99
  * 12 mg for patients 3-8.99 years of age
  * 15 mg for patients >9 years of age
  In Treatment Course 3:
  Intrathecally on day 1 at the age-defined dose
  Other Names: Otrexup; Rasuvo; Rheumatrex; Trexall; Amethopterin; Methotrexate Sodium; MTX
Drug: Cyclophosphamide — Course 2 only: • 1000mg/m2/day IV over 30 minutes to be given on day 1.
  Other Names: Cytoxan; Neosar
Drug: 6-thioguanine — Treatment Course 2 only: • 60 mg/m2/day to be given orally on days 1 through 14.
  Other Names: Thioguanine Tabloid; 6-TG; 2-Amino-6-Mercaptopurine

SUMMARY:
This is a phase I/II study of an investigational drug called ABT-751, produced by Abbott Laboratories, given in combination with chemotherapy drugs used to treat acute lymphoblastic leukemia (ALL) that has come back (recurred). The phase I portion of this study is being done to find the highest dose of ABT-751 that can be given safely in combination with other chemotherapy drugs. A safe dose is one that does not result in unacceptable side effects. After a safe dose for ABT-751 given with chemotherapy has been found, the study will add additional patients to find out if ABT-751 (given at the maximal safe dose) when given with additional chemotherapy is an effective therapy for the treatment of children with relapsed ALL. It is expected that approximately 15-35 children and young adults will take part in this study.

DETAILED DESCRIPTION:
All patients will receive the 2 courses of chemotherapy unless medical complications prevent the administration of some of the drugs. Treatment for the first 2 courses of therapy will last about 2 months.

Treatment on this study will consist of a combination of 8 anti-cancer medications. The 8 anticancer medicines are ABT-751, dexamethasone, PEG-asparaginase, doxorubicin, cytarabine (Ara-C), methotrexate (MTX), cyclophosphamide, and 6-thioguanine. All the drugs except ABT-751 are well known anti-cancer drugs and have been used extensively in the treatment of cancer.

During the Phase I portion of this study, when you enroll, you will be given an assigned dose of ABT-751. The dose of ABT-751 will be based on doses given in previous studies done with adults and children. At each dose level of ABT-751, between 3 and 6 children will receive ABT-751 in combination with chemotherapy. If the side effects are not too severe, the next group of children will receive a higher dose. The dose will continue to be increased until we find the dose that causes serious side effects. Your dose of ABT-751 will not be increased. If you have bad side effects, your dose may be decreased.

The dose used during the Phase 2 part of this study will be determined by the outcome of the Phase I study. The highest dose used in Phase I that was tolerated without serious side effects will be the one used in Phase 2.

ELIGIBILITY:
Inclusion Criteria

1. Age Patients must be < 21 years of age when enrolled onto this study. T2005-001 Protocol version 6/27/2007 17
2. Diagnosis

   Patients must have relapsed or refractory ALL with a M3 marrow (marrow blasts >25%) without clinical evidence of testicular disease or laboratory evidence of CNS disease defined as CSF WBC > 5 cells/microliter and blasts. (See Appendix I for method of evaluating traumatic lumbar punctures.) Patients in early first relapse (defined as a patient who relapses less than 36 months from their initial remission [CR1]) are eligible for the phase I portion of the trial.
3. Performance Level Karnofsky > 60% for patients > 10 years of age and Lansky > 60% for patients < 10 years of age.
4. Prior Therapy Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

   1. Prior anthracycline exposure: Patients must have less than 300mg/m2 lifetime exposure of anthracycline chemotherapy. (See Appendix III for calculation criteria)
   2. Stem Cell Transplant (SCT): Patients are eligible 6 months after allogeneic stem cell transplant as long as patients are not actively being treated for graft-versus-host-disease (GvHD).
   3. During the phase I portion of the trial, there is no limit on the number of prior treatment regimens.
   4. During the phase II portion of the trial, patients must have had two or more prior therapeutic attempts defined as:

      * Persistent initial disease after two induction attempts, or
      * Relapse after one-reinduction attempt (2nd relapse), or
      * Persistent disease after first relapse and initial re-induction attempt (Patients in any first relapse are not eligible for the phase II portion of the study)
   5. During the phase II portion of the trial, patients must have no more than 3 prior therapeutic attempts and it must be at least 6 months since the last treatment with a "VPLD" induction/re-induction regimen.
5. Reproductive Function

   1. Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed prior to enrollment and within 48 hours of starting therapy.
   2. Female patients with infants must agree not to breastfeed their infants while on this study.
   3. Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study and for 3 months following completion of therapy.

Exclusion Criteria

1. Drug Allergies

   Patients will be excluded if they have allergies to the following drugs:
   * Asparaginase products
   * Sulfa containing medications
2. Renal Function Patients will be excluded if their serum creatinine is > the upper limit of normal (ULN) for age at the institution's laboratory.
3. Liver/Pancreatic Function

   1. Direct bilirubin > 1.5x the institutional ULN for age. A total bilirubin result that is less than 1.5 times the institutional ULN for age may be used for eligibility if a direct bilirubin result is not available.
   2. SGPT (ALT) > 4 x institutional ULN
   3. Grade 3 or greater pancreatitis as defined by the CTCAE v3.0
   4. Amylase or Lipase > 2 x institutional ULN
4. Cardiac Function Patients will be excluded if their shortening fraction by echocardiogram is less than 30%.
5. Infection Patients will be excluded if they have an active, uncontrolled infection.

   1. Patients with grade 2 or greater motor or sensory neuropathy per CTC 3.0 criteria.
   2. Patients with grade 2 or greater Ileus (neuroconstipation) per CTC 3.0 criteria.
   3. Patients currently being treated with coumadin.
   4. Patients currently being treated with colchicines.
   5. Patients planning on receiving other investigational agents while on this study. (An investigational agent is defined as any drug not currently approved for use in humans.)
   6. Patients planning on receiving other anti-cancer therapies while on this study.
   7. Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
   8. Patients who, based on BSA and current dose level, require a daily dose of ABT-751 that is less than 25mg per day.
   9. Patients who have started protocol therapy prior to enrollment. Patient may still enroll if IT Ara-C or IT MTX were given within 48 hours of study enrollment as part of the diagnostic lumbar procedure. These patients will not participate in the CSF PK portion of the study.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2006-05-22; Primary Completion 2009-05-19 (Actual); Study Completion 2009-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Gaynon, MD, Study Chair — Childrens Hospital Los Angeles, Therapeutic Advances in Childhood Leukemia Consortium
Locations (5):
- United States (5):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - UCSF School of Medicine, San Francisco, California
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- See also: Therapeutic Advances in Childhood Leukemia & Lymphoma Consortium web site — http://www.tacl.us

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Starting dose for study is 80 mg/m2/day of ABT-751
- Dose Level 0: De-escalation dose due to DLTs: 65 mg/m2/day of ABT-751
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 0
Started | 5 | 4
Treatment Course 1 | 5 | 3
Treatment Course 2 | 1 | 1
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 0 | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 3 | 7
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Experienced Dose Limiting Toxicity From ABT-751
Description: ABT-751 was given daily for 21 days for a period of 28 day course in combination with dexamethasone, PEG-asparaginase, and doxorubicin. The occurrence of a dose limiting toxicity (DLT) was evaluated at the end of the 28 day course.
  DLT will be defined as any of the following events that are deemed by the investigator as probably or definitely attributable to ABT-751. Toxicity grade follows the CTCAE criteria, version 3.0. A copy of the CTCAE can be downloaded from the CTEP home page (http://ctep.cancer.gov).
  * Grade 3 or 4 Ileus
  * Grade 3 or 4 Constipation
  * Grade 3 or 4 Gastrointestinal obstruction, any location
  * Grade 3 or 4 Sensory Neuropathy
  * Grade 3 or 4 Motor Neuropathy
  * Grade 3 or 4 Neuropathic pain lasting longer than 24 hours despite medical intervention
  * Grade 3 or 4 Hypoxia in the absence of anemia or infection
  * Grade 4 Alanine aminotransferase (ALT) which does not return to
Time Frame: Each dose level is evaluated
Population: Number of participants that completed at least 1 course of treatment and are evaluable for toxicities.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 0
Number analyzed (Participants) | 5 | 4
Participants
  # of patients with DLT | 2 | 0
  # of patients without DLT | 3 | 4

2. Primary Outcome: Number of Patients That Achieved Complete Response to ABT-751
Description: Complete response (CR) is the occurrence of all of the following on approximately Day 29: less than 5% leukemic blasts in the bone marrow aspirate with no evidence of leukemic blasts in the CSF or peripheral blood and recovery of peripheral blood counts of an Absolute neutrophil count (ANC) > 750/μL and Platelet count > 75,000 μL.
Time Frame: Day 29 of Course 1
Population: Number of patients that completed at least 1 course of treatment and was evaluable for response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 0
Number analyzed (Participants) | 5 | 4
Participants
  # of patients not achieving complete response | 4 | 1
  # of patients who achieved complete response | 1 | 3

3. Secondary Outcome: Number of Patients With Occurrence of Toxic Death
Description: The occurrence of toxic death at anytime that is definitely, probably or possibly related to the treatment.
Time Frame: From the first dose of study therapy until 30 days after last therapy dose. Last dose protocol therapy is on day 21.
Population: Number of patients that completed at least 1 course of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 0
Number analyzed (Participants) | 5 | 4
Participants
  # of patients that experienced toxic death | 0 | 0
  # of patients that did not experience toxic death | 5 | 4

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events will be collected and reported on the electronic case report forms beginning with the first dose of investigational product until 30 days following the last dose of ABT-751, whether elicited or spontaneously reported by the patient, up to day 51 days (30 days after day 21, last day of the protocol therapy).
Description: The definition of adverse event (AE) and serious adverse event (SAE) do not differ from the clinicaltrials.gov definitions
Arm/Group | Dose Level 1 | Dose Level 0
All-Cause Mortality (participants affected / at risk) | 4/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 5/5 | 4/4
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=5) | Dose Level 0 (N=4)
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dehydration (Gastrointestinal disorders) | 1 | 0
Diarrhea NOS (Gastrointestinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3
Hyperglycemia NOS (Metabolism and nutrition disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Infection w/ Gr 3/4 ANC, Blood (Infections and infestations) | 4 | 1
Infection w/ Gr 3/4 ANC, Nose (Infections and infestations) | 1 | 0
Infection w/ Gr 3/4 ANC, Skin (Infections and infestations) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=5) | Dose Level 0 (N=4)
Abdominal distention (General disorders) | 1 | 0
Abdominal pain NOS (General disorders) | 2 | 3
Activated partial thromboplastin time prolonged (Blood and lymphatic system disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 5 | 4
Alkalosis NOS (Metabolism and nutrition disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 2
Blood bicarbonate decreased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Blood fibrinogen (Investigations) | 1 | 1
Blood/Bone Marrow-Other (Blood and lymphatic system disorders) | 5 | 4
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Caecitis (Gastrointestinal disorders) | 1 | 0
Cardiac-Other (Cardiac disorders) | 2 | 1
Clostridial infection NOS (Infections and infestations) | 1 | 0
Colitis NOS (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Diarrhea NOS (Gastrointestinal disorders) | 3 | 2
Dizziness (Nervous system disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Dyspepsia Heartburn (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Dermatology - Other (Skin and subcutaneous tissue disorders) | 1 | 0
Edema - limb (General disorders) | 1 | 0
Epistaxis (Vascular disorders) | 2 | 0
Fatigue (General disorders) | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Gastro-Other (Gastrointestinal disorders) | 1 | 0
Haemoglobin (Blood and lymphatic system disorders) | 4 | 4
Headache (Nervous system disorders) | 5 | 4
Hepatic infection (Hepatobiliary disorders) | 1 | 0
Hepatobiliary/Pancreas-Other (Hepatobiliary disorders) | 1 | 0
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia NOS (Metabolism and nutrition disorders) | 3 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 2
Hypernatremia (Metabolism and nutrition disorders) | 1 | 1
Hypertension NOS (Vascular disorders) | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 3
Hypoglycemia NOS (Metabolism and nutrition disorders) | 2 | 3
Hypokalemia (Metabolism and nutrition disorders) | 3 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 1
Hypotension NOS (Vascular disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Ileus paralytic (Gastrointestinal disorders) | 4 | 4
Infection w/ Gr 3/4 ANC, Blood (Infections and infestations) | 1 | 0
Infection w/ Gr 3/4 ANC, Urinary tract NOS (Infections and infestations) | 1 | 0
Infection w/ unk ANC, Urinary tract NOS (Infections and infestations) | 1 | 0
Left ventricular failure (Cardiac disorders) | 5 | 4
Leukopenia NOS (Blood and lymphatic system disorders) | 2 | 2
Metabolic/Lab-Other (Metabolism and nutrition disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Neuralgia NOS (Nervous system disorders) | 5 | 4
Neurology - Other (Nervous system disorders) | 1 | 0
Neutrophil count (Blood and lymphatic system disorders) | 2 | 2
Oral pain (General disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain NOS (General disorders) | 1 | 0
Pain-Other (General disorders) | 2 | 2
Peripheral motor neuropathy (Nervous system disorders) | 5 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 4
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Platelet count decreased (Blood and lymphatic system disorders) | 3 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Pulmonary-Other (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pyrexia (General disorders) | 0 | 1
Radiation mucositis (Injury, poisoning and procedural complications) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Respiratory tract infection NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rigors (General disorders) | 2 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Vomiting NOS (Gastrointestinal disorders) | 3 | 3
Weight decreased (Metabolism and nutrition disorders) | 3 | 1

LIMITATIONS AND CAVEATS:
Study was terminated early due to lack of accrual. Data were not analyzed for outcome variables.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days